CLINICAL TRIAL: NCT00850876
Title: Randomized Cross-over Trials of the Effect of Heated Humidified CPAP Versus Non-humidified CPAP on Nasal Physiology
Brief Title: Heated Humidified Continuous Positive Airway Pressure and Nasal Physiology
Status: Completed | Type: Observational
Sponsor: University of Athens (Other)
Responsible Party: Ioannis Koutsourelakis, 1Center of Sleep Disorders Medical School of Athens University, Department of Critical Care and Pulmonary Services
Other Study IDs: UOA-12008
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Last update posted 2010-04-09 (Estimated); Status verified 2010-04

CONDITIONS: Obstructive Sleep Apnea Syndrome; Nasal Obstruction
MeSH Terms: conditions — Sleep Apnea, Obstructive; Nasal Obstruction

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Nasal wash will be performed using a technique adapted by Hurst et al. Briefly, a 12-French Foley catheter (Bard, Crawley, UK), modified by removal of the tip distal to the balloon, was inserted into the nostril and inflated with sufficient air to form a comfortable seal (typically 7-10ml). With the patients head flexed 45o forward, 7ml of warmed 0.9% saline will be instilled through the catheter and washed in and out of the nasal cavity three times. A portion of the pooled wash from both nostrils will be centrifuged to yield a supernatant for analysis of inflammatory cytokines (IL-6, IL-8, TNF-a, IL-10).
Oversight: Data Monitoring Committee: No

SUMMARY:
Nasal continuous positive airway pressure can cause nasal side effects which can compromise compliance to therapy. Humidifiers can attenuate this effect. However, the mechanism by which humidified CPAP alleviates nasal symptoms has never been assessed objectively in OSA patients. Therefore, the purpose of this study is to examine the effect of humidified CPAP on nasal airway physiology with combined measurements of nasal resistance and level of inflammatory markers. The investigators' hypothesis is that the addition of heated humidification in CPAP decreases nasal airway resistance and nasal mucosal inflammation markers and thus, ameliorates nasal symptoms of OSAS patients.

DETAILED DESCRIPTION:
Introduction-Rationale:

Nasal continuous positive airway pressure (CPAP) is considered to be the "gold standard" of obstructive sleep apnoea (OSA) treatment [1]. The most common side effects are nasal congestion, stuffiness or dryness and rhinorrhea which have been reported in up to 68% of patients responding to a questionnaire about nasal CPAP. In many of them, CPAP compliance is accordingly compromised.

The mechanisms by which CPAP provokes nasal symptoms have been thoroughly studied only in healthy volunteers and a rodent model. Indeed, Richards et al demonstrated that mouth leaks causing high unidirectional nasal airflow increased nasal airway resistance and this response could be largely prevented by heated humidification of the inspired air. Similarly, Togias et al showed an elevated release of inflammatory mediators (histamine, prostaglandin D2, kinins) in nasal wash fluids when compressed cold and dry air was delivered through the nose. This effect was also prevented when warm and moist air was delivered. More recently, Almendros et al provided evidence that CPAP use in rats triggered early nasal inflammation.

Of the variety of methods used to treat nasal symptoms during CPAP treatment, the most common is humidification of the inspired air. However, the mechanism Oby which humidified CPAP attenuates nasal symptoms has never been assessed objectively in OSA patients. Therefore, the purpose of this study is to examine the effect of humidified CPAP on nasal airway physiology with combined measurements of nasal resistance and level of inflammatory markers. Our hypothesis is that the addition of heated humidification in CPAP decreases nasal airway resistance and nasal mucosal inflammation markers and thus, ameliorates nasal symptoms of OSAS patients.

Study design:

BASELINE: 1. NASAL SYMPTOMS 2. NASAL RESISTANCE 3. NASAL WASH (IL-6, IL-8, TNF-a, IL-10)

3 weeks humidified CPAP --------------> 3 weeks non-humidified CPAP <--------------

AFTER TREATMENT: 1. NASAL SYMPTOMS 2. NASAL RESISTANCE 3. NASAL WASH (IL-6, IL-8, TNF-a, IL-10)

Methods:

1. Nasal symptoms will be assessed using a five point Nasal Score. Each of the five principal nasal symptoms of rhinorrhoea, post-nasal drip, sneezing, impaired sense of smell and nasal blockage will be binary coded as present/increased over baseline (1) or absent/not (0) and summed to yield a total Nasal Score between zero and five.
2. Nasal resistance will be assessed by active anterior and posterior rhinomanometry in both seated and supine (for 10 min) positions.
3. Nasal wash will be performed using a technique adapted by Hurst et al. Briefly, a 12-French Foley catheter (Bard, Crawley, UK), modified by removal of the tip distal to the balloon, was inserted into the nostril and inflated with sufficient air to form a comfortable seal (typically 7-10ml). With the patients head flexed 45o forward, 7ml of warmed 0.9% saline will be instilled through the catheter and washed in and out of the nasal cavity three times. A portion of the pooled wash from both nostrils will be centrifuged to yield a supernatant for analysis of inflammatory cytokines.

By this protocol, the following are expected: a) the reason for potential congestion and inflammatory response is cold and dry air passing through the nostrils (mechanical irritation cannot be the reason, as the pressure is equivalent in both sessions), and b) heated and humidified CPAP prevents (and not treats) nasal congestion.

ELIGIBILITY:
Inclusion Criteria:

1. Obstructive sleep apnea syndrome defined as apnea/hypopnoea index greater than 20,
2. Initiation of continuous positive airway pressure, and
3. Symptomatic nasal obstruction.

Exclusion Criteria:

1. No medication known to influence nasal resistance (antihistamines, vasoconstrictors, vasodilators, topical or systemic steroids, and recreation drugs),
2. No smoking,
3. No upper or lower respiratory tract disease (e.g. upper respiratory tract infection, rhinitis, sinusitis, chronic obstructive pulmonary disease), including a history of nasal allergy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who refer to the Center of Sleep Disorders of "Evangelismos" General Hospital of Athens for suspected sleep disordered breathing.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-09; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Koutsourelakis, MD, Principal Investigator — 1Center of Sleep Disorders Medical School of Athens University, Department of Critical Care and Pulmonary Services
Locations (1):
- Department of Critical Care and Pulmonary Services, Evangelismos Hospital, Athens, Greece

REFERENCES:
- [Background] Kushida CA, Chediak A, Berry RB, Brown LK, Gozal D, Iber C, Parthasarathy S, Quan SF, Rowley JA; Positive Airway Pressure Titration Task Force; American Academy of Sleep Medicine. Clinical guidelines for the manual titration of positive airway pressure in patients with obstructive sleep apnea. J Clin Sleep Med. 2008 Apr 15;4(2):157-71. PMID 18468315
- [Background] Willing S, San Pedro M, Driver HS, Munt P, Fitzpatrick MF. The acute impact of continuous positive airway pressure on nasal resistance: a randomized controlled comparison. J Appl Physiol (1985). 2007 Mar;102(3):1214-9. doi: 10.1152/japplphysiol.00639.2006. Epub 2006 Dec 7. PMID 17158250
- [Background] Randerath WJ, Meier J, Genger H, Domanski U, Ruhle KH. Efficiency of cold passover and heated humidification under continuous positive airway pressure. Eur Respir J. 2002 Jul;20(1):183-6. doi: 10.1183/09031936.02.00267902. PMID 12166568
- [Background] Mador MJ, Krauza M, Pervez A, Pierce D, Braun M. Effect of heated humidification on compliance and quality of life in patients with sleep apnea using nasal continuous positive airway pressure. Chest. 2005 Oct;128(4):2151-8. doi: 10.1378/chest.128.4.2151. PMID 16236868
- [Background] Bossi R, Piatti G, Roma E, Ambrosetti U. Effects of long-term nasal continuous positive airway pressure therapy on morphology, function, and mucociliary clearance of nasal epithelium in patients with obstructive sleep apnea syndrome. Laryngoscope. 2004 Aug;114(8):1431-4. doi: 10.1097/00005537-200408000-00022. PMID 15280722
- [Background] Hurst JR, Perera WR, Wilkinson TM, Donaldson GC, Wedzicha JA. Systemic and upper and lower airway inflammation at exacerbation of chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2006 Jan 1;173(1):71-8. doi: 10.1164/rccm.200505-704OC. Epub 2005 Sep 22. PMID 16179639
- [Background] Richards GN, Cistulli PA, Ungar RG, Berthon-Jones M, Sullivan CE. Mouth leak with nasal continuous positive airway pressure increases nasal airway resistance. Am J Respir Crit Care Med. 1996 Jul;154(1):182-6. doi: 10.1164/ajrccm.154.1.8680678.
- [Background] Togias AG, Naclerio RM, Proud D, Fish JE, Adkinson NF Jr, Kagey-Sobotka A, Norman PS, Lichtenstein LM. Nasal challenge with cold, dry air results in release of inflammatory mediators. Possible mast cell involvement. J Clin Invest. 1985 Oct;76(4):1375-81. doi: 10.1172/JCI112113. PMID 2414318
- [Background] Almendros I, Acerbi I, Vilaseca I, Montserrat JM, Navajas D, Farre R. Continuous positive airway pressure (CPAP) induces early nasal inflammation. Sleep. 2008 Jan;31(1):127-31. doi: 10.1093/sleep/31.1.127. PMID 18220086
- [Derived] Koutsourelakis I, Vagiakis E, Perraki E, Karatza M, Magkou C, Kopaka M, Roussos C, Zakynthinos S. Nasal inflammation in sleep apnoea patients using CPAP and effect of heated humidification. Eur Respir J. 2011 Mar;37(3):587-94. doi: 10.1183/09031936.00036910. Epub 2010 Jul 1. PMID 20595158